CLINICAL TRIAL: NCT02080468
Title: A Phase 1, Open-Label, Randomized, 2-Arm Study to Evaluate the Effect of Ethinyl Estradiol/Norgestimate (Ortho Cyclen®), a Weak CYP3A4 Inhibitor, on the Pharmacokinetics of Lomitapide in Healthy Female Subjects
Brief Title: Evaluate the Effect of Ethinyl Estradiol/Norgestimate on the Pharmacokinetics of Lomitapide in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AEGR-733-029
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Effect; Ethinyl Estradiol/Norgestimate; Pharmacokinetics; Lomitapide.
MeSH Terms: interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Lomitapide & EE/Norgestimate - Taken Together (Experimental): Lomitapide & EE/Norgestimate - Taken Together 2 single oral doses of lomitapide (20 mg) (Day 1 & Day 22) 21 single oral doses of EE/Norgestimate(Day 8 through day 28)
  Interventions: Drug: lomitapide; Drug: EE/norgestimate
- Arm 2: Lomitapide & EE/Norgestimate - Taken 12 Hours Apart (Experimental): Lomitapide & EE/Norgestimate - Taken 12 hours apart 2 single oral doses of lomitapide (20 mg) (Day 1 & Day 22) 21 single oral doses of EE/Norgestimate(Day 9 through day 29)
  Interventions: Drug: lomitapide; Drug: EE/norgestimate

INTERVENTIONS:
Drug: lomitapide — 20 mg
  Other Names: Juxtapid
Drug: EE/norgestimate — 1x0.035-mg EE/0.25-mg norgestimate tablet
  Other Names: Ortho Cylclen

SUMMARY:
The primary objective of this study is to assess the effect of ethinyl estradiol (EE)/norgestimate, a weak cytochrome P450 (CYP) 3A4 inhibitor, on the pharmacokinetics (PK) of lomitapide and 2 primary metabolites, M1 and M3.

DETAILED DESCRIPTION:
This study will be a single center, randomized, open-label, 2 arm study to evaluate the effects of EE/norgestimate, a weak CYP3A4 inhibitor, on the PK of lomitapide in healthy female subjects when EE/norgestimate is administered simultaneously with lomitapide and when administration is separated by 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females, between 18 and 40 years of age inclusive
2. BMI between 18.5 and 30.0 kg/m2, inclusive; total body weight of >110 lbs (50 kg);
3. in good health, determined by no clinically significant or relevant abnormalities identified by a detailed medical history and physical exam
4. no known history of hypersensitivity or previous intolerance to lomitapide or EE/norgestimate
5. creatine phosphokinase, AST, and ALT levels must be below 1.5 times the upper limit of normal
6. clinical laboratory evaluations within the reference range for the test laboratory
7. negative test for selected drugs of abuse
8. negative hepatitis panel and negative HIV antibody screens
9. are of childbearing potential(ie, not postmenopausal or surgically sterile). All subjects must have a negative serum beta pregnancy test.
10. able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

1. significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disorder
2. history of unexplained breast abnormalities or abnormal uterine bleeding
3. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
4. history of stomach or intestinal surgery or resection
5. history of Gilbert's Syndrome or suspicion of Gilbert's Syndrome
6. subjects who have an abnormality in the 12-lead ECG
7. use of any drugs of abuse for 6 months prior to Check-in;
8. subjects who consume more than 14 units of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse within 1 year prior to Check-in
9. use of any tobacco- or nicotine-containing products within 6 months prior to Check-in;
10. participation in any other investigational study drug trial within 30 days prior to Check-in;
11. use of any prescription medications/products within 14 days prior to Check-in unless deemed acceptable by the Investigator and Sponsor
12. use of any over-the-counter, nonprescription preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator and Sponsor
13. use of alcohol-, grapefruit- (including star fruit), or caffeine-containing foods or beverages within 72 hours prior to Check-in and through Study Completion
14. use of oral (except scheduled administration of EE/norgestimate), implantable, injectable, or transdermal contraceptives
15. use of hormone replacement therapy
16. poor peripheral venous access;
17. donation of blood (500 mL) from 30 days prior to Screening through Study Completion
18. receipt of blood products within 2 months prior to Check-in;
19. any acute or chronic condition, scheduled hospitalization (inclusive of elective surgery during study) or scheduled travel prior to completion of all study procedures which, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study;
20. subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2014-04-24 (Actual); Study Completion 2014-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sumeray, MD, Study Chair — Cheif Medical Officer; T. Alex King, MD, CPI, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lomitapide & EE/Norgestimate - Taken Together: 2 single oral doses of lomitapide (20 mg) (Day 1 & Day 22)
  21 single oral doses of EE/Norgestimate(Day 8 through day 28)
  lomitapide: 20 mg
  EE/norgestimate: 1x0.035-mg EE/0.25-mg norgestimate tablet
- Lomitapide & EE/Norgestimate - Taken 12 Hours Apart: 2 single oral doses of lomitapide (20 mg) (Day 1 & Day 22)
  21 single oral doses of EE/Norgestimate(Day 9 through day 29)
  lomitapide: 20 mg
  EE/norgestimate: 1x0.035-mg EE/0.25-mg norgestimate tablet
Period: Overall Study
Arm/Group | Lomitapide & EE/Norgestimate - Taken Together | Lomitapide & EE/Norgestimate - Taken 12 Hours Apart
Started | 16 | 16
Completed | 14 | 14
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lomitapide & EE/Norgestimate - Taken Together | Lomitapide & EE/Norgestimate - Taken 12 Hours Apart | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.4) | 29 (5.7) | 29 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Arm 1 (Lomitapide & EE/Noregestimate - Taken Together)
Description: Maximum observed plasma concentration of lomitapide and its 2 primary metabolites, M1 & M3
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: The Pharmacokinetic Analysis population included all subjects. Only subjects who completed both periods were included in the ANOVA analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK of Lomitapide (Lomitapide Alone): PK of lomitapide following administration of lomitapide alone
- PK of Lomitapide (Coadministered Simultaneously): PK of lomitapide following administration of lomitapide coadministered with EE/Norgestimate simultaneously
- PK of M1 (Lomitapide Alone): PK of M1 following administration of lomitapide alone
- PK of M1 (Coadministered Simultaneously): PK of M1 following administration of lomitapide coadministered with EE/Norgestimate simultaneously
- PK of M3 (Lomitapide Alone): PK of M3 following administration of lomitapide alone
- PK of M3 (Coadministered Simultaneously): PK of M3 following administration of lomitapide coadministered with EE/Norgestimate simultaneously
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng/mL | 1.03 (39.1) | 1.39 (58.4) | 2.96 (27.0) | 2.95 (19.4) | 36.3 (32.1) | 34.0 (27.9)

2. Primary Outcome: Tmax for Arm 1 (Lomitapide & EE/Noregestimate - Taken Together)
Description: Time to reach maximum observed plasma concentration of lomitapide and its 2 primary metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
hr | 6.00 [4.00 to 12.0] | 5.00 [1.00 to 18.0] | 8.28 [5.00 to 12.0] | 6.00 [2.00 to 12.0] | 5.02 [3.00 to 12.0] | 3.97 [1.00 to 6.00]

3. Primary Outcome: AUC0-t for Arm 1 (Lomitapide & EE/Noregestimate - Taken Together)
Description: Area under the concentration-time curve from zero to last quantifiable concentration of lomitapide and its 2 primary metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng*hr/mL | 33.5 (35.0) | 42.7 (49.5) | 89.3 (35.6) | 96.8 (32.1) | 456 (41.2) | 371 (36.1)

4. Primary Outcome: AUC0-∞ for Arm 1 (Lomitapide & EE/Noregestimate - Taken Together)
Description: Area under the concentration-time curve from zero to infinity of lomitapide and its 2 primary metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng*hr/mL | 36.5 (34.8) | 46.5 (49.1) | 91.4 (35.8) | 99.4 (32.4) | 463 (40.9) | 377 (36.0)

5. Primary Outcome: t1/2 for Arm 1 (Lomitapide & EE/Noregestimate - Taken Together)
Description: Apparent terminal elimination half-life of lomitapide and its 2 primary metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Coadministered Simultaneously) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered Simultaneously) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered Simultaneously)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
hr | 51.0 (16.1) | 53.6 (19.0) | 32.5 (20.3) | 36.8 (30.3) | 38.3 (32.7) | 39.8 (26.2)

6. Secondary Outcome: Cmax for Arm 2 (Lomitapide & EE/Noregestimate - 12 Hours Apart)
Description: Maximum observed plasma concentration of lomitapide and its metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- PK of Lomitapide (Codministered 12 Hours Apart): PK of lomitapide following administration of lomitapide coadministered with EE/Norgestimate 12 hours apart
- PK of M1 (Coadministered 12 Hours Apart): PK of M1 following administration of lomitapide coadministered with EE/Norgestimate 12 hours apart
- PK of M3 (Coadministered 12 Hours Apart): PK of M3 following administration of lomitapide coadministered with EE/Norgestimate 12 hours apart
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Codministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng/mL | 1.05 (50.7) | 1.39 (56.5) | 2.87 (20.6) | 3.04 (22.8) | 37.8 (26.2) | 33.0 (28.0)

7. Secondary Outcome: Tmax for Arm 2 (Lomitapide & EE/Noregestimate - 12 Hours Apart)
Description: Time to reach maximum observed plasma concentration of lomitapide and its metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Mean (Full Range); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Codministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
hr | 8.00 [5.00 to 10.0] | 8.00 [3.00 to 11.8] | 9.07 [5.00 to 12.0] | 8.00 [3.00 to 11.9] | 6.00 [5.00 to 10.0] | 5.50 [2.00 to 8.40]

8. Secondary Outcome: AUC0-t for Arm 2 (Lomitapide & EE/Noregestimate - 12 Hours Apart)
Description: Area under the concentration-time curve from zero to last quantifiable concentration of lomitapide and its metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Codministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng*hr/mL | 37.6 (49.9) | 46.5 (55.1) | 92.3 (31.1) | 93.7 (34.2) | 520 (30.1) | 377 (31.9)

9. Secondary Outcome: AUC0-∞ for Arm 2 (Lomitapide & EE/Noregestimate - 12 Hours Apart)
Description: Area under the concentration-time curve from zero to infinity of lomitapide and its metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Codministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
ng*hr/mL | 41.1 (50.9) | 51.2 (55.3) | 94.5 (31.3) | 96.4 (34.6) | 528 (30.0) | 383 (31.7)

10. Secondary Outcome: t1/2 for Arm 2 (Lomitapide & EE/Noregestimate - 12 Hours Apart)
Description: Apparent terminal elimination half-life of lomitapide and its metabolites, M1 & M3.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 169 hours after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | PK of Lomitapide (Lomitapide Alone) | PK of Lomitapide (Codministered 12 Hours Apart) | PK of M1 (Lomitapide Alone) | PK of M1 (Coadministered 12 Hours Apart) | PK of M3 (Lomitapide Alone) | PK of M3 (Coadministered 12 Hours Apart)
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 16 | 14
hr | 51.0 (22.2) | 52.0 (16.1) | 36.2 (21.0) | 37.2 (19.1) | 38.0 (28.0) | 33.6 (23.2)

ADVERSE EVENTS:
Arm/Group | Lomitapide & EE/Norgestimate - Taken Together | Lomitapide & EE/Norgestimate - Taken 12 Hours Apart
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 8/16 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomitapide & EE/Norgestimate - Taken Together (N=16) | Lomitapide & EE/Norgestimate - Taken 12 Hours Apart (N=16)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Vomitting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vessel Punction Site Pain (General disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in site contract